CLINICAL TRIAL: NCT05893927
Title: Evaluating the Clinical Impact of a PCP Developed Diabetes Education Mobile Web Application on Patients With Uncontrolled Type 2 Diabetes
Brief Title: Impact of a Diabetes Education Mobile Web Application on Patients With Uncontrolled Type 2 Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Reading Hospital and Medical Center (Other)
Collaborators: Reading Hospital Foundation (Unknown); Complete Statistical Services (Consult-Stat) (Unknown)
Responsible Party: Principal Investigator, Luis Murillo, Residency Faculty Associate, Director Hanna Center for Primary Care Research, The Reading Hospital and Medical Center
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-020
Record Dates: First submitted 2023-05-30; First posted 2023-06-08 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Diabetes Mellitus, Type 2; Diabetes Education; Lifestyle Modification
Keywords: Type 2 diabetes; Type II diabetes; uncontrolled type 2 diabetes; hyperglycemia; mobile web application; Diabetes education
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hyperglycemia

STUDY DESIGN:
Intervention Model Description: Participants will be recruited to participate in the study, and then randomized to one of two arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention arm (Experimental): Participants enrolled in the intervention arm will be given a 6-month access period to the diabetes education application designed by the study team. The web site will offer videos related to a specific areas of education concerning diabetes self-management. To encourage compliance, participant users will receive weekly notifications from the application that will guide them through viewing all videos in the series. Participants will continue routine follow-up appointments with their primary care physicians during the study period. There will be no restrictions on starting or stopping medications during the study period.
  Interventions: Other: Diabetes education web site application
- Control arm (No Intervention): Participants in the control arm will not have access to the Diabetes Application. They will continue follow-up appointments according to the standard of care with their primary care physician, diabetic educators, etc. There are no restrictions on starting or stopping medications for patients within the control arm.

INTERVENTIONS:
Other: Diabetes education web site application — The Diabetes education website application will contain informational videos for this protocol. The videos will include a welcome video and the categorical topics of Healthy Coping, Healthy Eating, Staying Active, Medications (Use and Safety), Problem Solving in Diabetes, and Disease Pathophysiology. Each category contains several videos providing education about a different component of diabetes care.
  Arms: Intervention arm

SUMMARY:
The goal of this clinical trial is to evaluate the use and effectiveness of a mobile web application (app) that is designed to educate and allow patients to manage diabetes and make sustainable lifestyle changes, and to study the impact of the app on clinical outcomes of diabetes (HA1C) and educational outcomes (Self-Efficacy for Diabetes Scale). The main question to answer is: Does the use of the Diabetes Application significantly affect clinical outcomes of diabetes and cardiometabolic risk factors (BMI and Blood Pressure)? Patients will be enrolled in one of two available arms of the study.

Participants in the 'intervention arm' will use the app to view educational information presented as videos in the following areas: Healthy Coping, Healthy Eating, Staying Active, Medications (Use and Safety), Problem Solving in Diabetes and Disease Pathophysiology. They will continue routine follow-up care with their primary care physicians during the study.

Participants in the 'control arm' will continue with their primary care physician in routine follow-up care, as normally scheduled.

Researchers will compare the intervention arm participants to the control arm participants to find out about and compare changes in HA1C, systolic blood pressure, diastolic blood pressure, and body mass index. Groups will also be compared on the basis of self-perceived confidence of managing their diabetes by way of the Diabetes Self Efficacy Scale.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of Type 2 Diabetes with HA1c >8.0
* Current patients of the Family Healthcare Center, Reading Hospital Tower health.

Exclusion Criteria:

* Identified special populations (pregnancy or individuals currently incarcerated)
* Patients without access to their own smart phone
* Any patient who is unable to provide their own informed consent to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin A1c | 6 months
  Blood Test
"Self-Efficacy for Diabetes Scale" | 6 months
  A validated (free to use) survey that examines self-perceived ability to manage diabetes. Scores are reported on a scale from 1-10. 1 reflecting Not at all confident and 10 reflecting confident. The minimum total value is 8, and the maximum value is 80. A higher score indicates that the individual has a better outcome, i.e., more confident that he/she can perform the task regularly at the present time.

SECONDARY OUTCOMES:
Body Mass Index | 6 months
  Height-to-weight ratio, an indicator of underweight, normal weight, or overweight/obese

CONTACTS AND LOCATIONS:
Overall Officials: Luis A Murillo, MD, MPH, Principal Investigator — Reading Hospital Tower Health
Locations (1):
- Reading Hospital, an affiliate of Tower Health, West Reading, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shan R, Sarkar S, Martin SS. Digital health technology and mobile devices for the management of diabetes mellitus: state of the art. Diabetologia. 2019 Jun;62(6):877-887. doi: 10.1007/s00125-019-4864-7. Epub 2019 Apr 8. PMID 30963188
- [Background] Ball E, Rivas C. Health Apps Require Co-development to Be Acceptable and Effective. Front Psychol. 2021 Jul 16;12:714453. doi: 10.3389/fpsyg.2021.714453. eCollection 2021. No abstract available. PMID 34335428
- [Background] Kao CK, Liebovitz DM. Consumer Mobile Health Apps: Current State, Barriers, and Future Directions. PM R. 2017 May;9(5S):S106-S115. doi: 10.1016/j.pmrj.2017.02.018. PMID 28527495
- [Background] Doyle-Delgado K, Chamberlain JJ. Use of Diabetes-Related Applications and Digital Health Tools by People With Diabetes and Their Health Care Providers. Clin Diabetes. 2020 Dec;38(5):449-461. doi: 10.2337/cd20-0046. PMID 33384470
- [Background] Ye Q, Khan U, Boren SA, Simoes EJ, Kim MS. An Analysis of Diabetes Mobile Applications Features Compared to AADE7: Addressing Self-Management Behaviors in People With Diabetes. J Diabetes Sci Technol. 2018 Jul;12(4):808-816. doi: 10.1177/1932296818754907. Epub 2018 Feb 1. PMID 29390917
- [Background] Bonoto BC, de Araujo VE, Godoi IP, de Lemos LL, Godman B, Bennie M, Diniz LM, Junior AA. Efficacy of Mobile Apps to Support the Care of Patients With Diabetes Mellitus: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. JMIR Mhealth Uhealth. 2017 Mar 1;5(3):e4. doi: 10.2196/mhealth.6309. PMID 28249834
- [Background] American Diabetes Association. 6. Glycemic Targets: Standards of Medical Care in Diabetes-2021. Diabetes Care. 2021 Jan;44(Suppl 1):S73-S84. doi: 10.2337/dc21-S006. PMID 33298417
- [Background] Cui M, Wu X, Mao J, Wang X, Nie M. T2DM Self-Management via Smartphone Applications: A Systematic Review and Meta-Analysis. PLoS One. 2016 Nov 18;11(11):e0166718. doi: 10.1371/journal.pone.0166718. eCollection 2016. PMID 27861583
- [Background] He Q, Zhao X, Wang Y, Xie Q, Cheng L. Effectiveness of smartphone application-based self-management interventions in patients with type 2 diabetes: A systematic review and meta-analysis of randomized controlled trials. J Adv Nurs. 2022 Feb;78(2):348-362. doi: 10.1111/jan.14993. Epub 2021 Jul 29. PMID 34324218
- [Background] Jeste DV, Palmer BW, Appelbaum PS, Golshan S, Glorioso D, Dunn LB, Kim K, Meeks T, Kraemer HC. A new brief instrument for assessing decisional capacity for clinical research. Arch Gen Psychiatry. 2007 Aug;64(8):966-74. doi: 10.1001/archpsyc.64.8.966. PMID 17679641
- [Background] Beckerle CM, Lavin MA. Association of Self-Efficacy and Self-Care With Glycemic Control in Diabetes. Diabetes Spectrum. 2013; 26(3): 172-178
- See also: Mobile Fact Sheet from Pew Research Center, published April 07, 2021 — https://www.pewresearch.org/internet/fact-sheet/mobile/